CLINICAL TRIAL: NCT01391104
Title: Reproducibility and Responsiveness of Exercise Tests in Pulmonary Arterial Hypertension
Brief Title: Responsiveness of Exercise Tests in Pulmonary Arterial Hypertension
Acronym: RESPONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Vincent Mainguy, Doctorant, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESPONS PAH
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Exercise; Six-minute walk test; sildenafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Motor Activity | interventions — Sildenafil Citrate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenalfil (Experimental): Patients will be assigned to sildenafil (20 mg tid) or placebo per os for 28 days in a randomized, double-blind manner. After a four-week wash-out period, patients will then be crossed over to the alternate therapy for the next 28 days.
  Interventions: Drug: Sildenafil
- Sugar Pill (Placebo Comparator): Patients will be assigned to sildenafil (20 mg tid) or placebo per os for 28 days in a randomized, double-blind manner. After a four-week wash-out period, patients will then be crossed over to the alternate therapy for the next 28 days.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Sildenafil — Sildenafil citrate is a phosphodiesterase type-5 inhibitor. Patients will be assigned to sildenafil (20 mg tid) or placebo per os for 28 days in a randomized, double-blind manner. After a four-week wash-out period, patients will then be crossed over to the alternate therapy for the next 28 days.
  Other Names: Revatio; Viagra
  Arms: Sildenalfil
Drug: Sugar Pill — Patients will be assigned to sildenafil (20 mg tid) or placebo per os for 28 days in a randomized, double-blind manner. After a four-week wash-out period, patients will then be crossed over to the alternate therapy for the next 28 days.
  Arms: Sugar Pill

SUMMARY:
Pulmonary arterial hypertension (PAH) is characterized by the progressive increase in pulmonary vascular resistance leading to shortness of breath and exercise intolerance. Exercise capacity has been used as the primary endpoint in most recent randomized controlled trials evaluating PAH-specific therapies as it correlates with functional class and survival in PAH. Exercise test is commonly assessed by the six-minute walk test (6MWT). However, there is commonly some discrepancy between significant clinical improvement and minor changes (generally <10% from baseline) in 6WMT following therapy. Because important clinical decisions are based on patients' functional capacity, a reproducible and sensitive exercise test is needed in PAH. The aim of this study was to compare the reproducibility and the responsiveness of the 6MWT, the endurance shuttle walk test (ESWT) and the cycle endurance test (CET) following pharmacological therapy in this disease.

ELIGIBILITY:
Inclusion Criteria:

* WHO functional class II or III
* Idiopathic PAH, familial PAH, or associated PAH due to connective tissue disease patients
* Mean pulmonary artery pressure ≥25 mmHg at rest
* Pulmonary capillary wedge pressure ≤15 mmHg

Exclusion Criteria:

* Prior use of phosphodiesterase type-5 inhibitors
* Unstable clinical condition over the last 4 months
* Recent syncope
* WHO functional class IV
* Left ventricular ejection fraction <40%
* Restrictive or obstructive lung disease
* Intrinsic musculoskeletal abnormality precluding exercise testing
* Patients with a pacemaker
* Treatment with systemic corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To compare the reproducibility and the responsiveness of the 6MWT, the endurance shuttle walk test (ESWT) and the cycle endurance test (CET) following pharmacological therapy in PAH. | 3 months
  After completing the 6MWT, the ESWT and the CET in a randomized order, patients will then be randomized to sildenafil (20mg tid) or placebo in a double-blind manner for 28 days. The three exercise tests will then be repeated. After a four-week of wash-out period, patients will repeat the three exercise test and then be crossed over to the alternate therapy for the next 28 days. The same experiments will be repeated after this period. The reproducibility of each exercise test will be assessed following placebo. The responsiveness of each exercise test will be assessed following sildenafil.

SECONDARY OUTCOMES:
To assess the efficacy of a combination therapy in pulmonary arterial hypertension (PAH). | 1 month
  Sildenafil will be added to the baseline therapy for one month (20mg tid). The efficacy of this combined therapy will be assessed by three different exercise tests and by a quality of life questionnaire.
To measure the physiological parameters induced by five different exercise tests in pulmonary arterial hypertension (PAH) | 2 weeks
  Within one week, PAH patients will performed five different exercise tests. During each test, a portable telemetric system (Oxycon, Jaegger, Germany) will be used to assess the respiratory cardiovascular adaptations. Symptoms of leg fatigue and dyspnea will be assessed using the Borg scale. Quadriceps fatigability will be assessed by volitional and non-volitional (twitch force, TWq) measurements of the quadriceps strength before and immediately after each test (Magstim Co. Ltd., Whitland, Dyfed, Wales, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, M.Sc., Principal Investigator — Laval University
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec (CRIUCPQ), Québec, Quebec, Canada